CLINICAL TRIAL: NCT01092026
Title: A Pilot Study to Assess the Feasibility of Unrelated Umbilical Cord Blood Transplantation With Coinfusion of Third-party Mesenchymal Stem Cells After Myeloablative or Nonmyeloablative Conditioning in Patients With Hematological Malignancies
Brief Title: Unrelated Umbilical Cord Blood Transplantation With Coinfusion of Mesenchymal Stem Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHS-UCB2009
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2018-05

CONDITIONS: Allogeneic Stem Cell Transplantation
MeSH Terms: interventions — Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Intervention Model Description: Patients will receive either myeloablative or reduced intensity conditioning. One or 2 cord blood transplants will be transplanted, followed by infusion of a third-party mesenchymal stem cell transplant
Oversight: Data Monitoring Committee: No

ARMS (1):
- cord blood transplant (Experimental): Eligible patients receive cord blood transplantation with coinfusion of mesenchymal stem cells
  Interventions: Other: cord blood transplantation

INTERVENTIONS:
Other: cord blood transplantation — One or two cord blood transplants with co-infusion of third-party mesenchymal stem cells after pre-transplant preparative regimen

SUMMARY:
A pilot study to assess the feasibility of unrelated umbilical cord blood transplantation with coinfusion of third-party mesenchymal stem cells after myeloablative or nonmyeloablative conditioning in patients with hematological malignancies.

This is a multicenter single arm, phase I-II pilot study. The primary objective of this study is to determine the feasibility of Umbilical Cord Blood (UCB) Hematopoietic Stem Cell Transplantation (HSCT) with co-infusion of third party mesenchymal stem cells as assessed by the treatment-related mortality at d100 after transplant.

Patient inclusion criteria:

Age 15-60 yrs, Patients for whom allogeneic stem cell transplantation is the preferred treatment option, with the following hematological malignancies: acute myeloid leukemia, acute lymphoblastic leukemia, high risk myelodysplastic syndrome, advanced lymphoproliferative disorders, chronic myeloid leukemia (refractory or intolerant to second-line tyrosine kinase inhibitors), multiple myeloma, Informed consent given, Patient exclusion criteria, Previous allogeneic transplant, Progressive malignant disease, Significant organ damage as a contraindication to allotransplantation, Significant psychiatric or neurological disorder, Uncontrolled viral, fungal or bacterial infection, Pregnancy, HIV positive, Patients will receive either myeloablative or reduced intensity conditioning. One or 2 cord blood transplants will be transplanted, followed by infusion of a third-party mesenchymal stem cell transplant, Adverse event reporting Belgian Hematology Society (BHS) transplant committee will establish a protocol review committee which will organize a central monitoring of the study. Within the context of allogeneic Hematopoietic Stem Cell Transplantation (HSCTx) many severe events are likely to occur.

Statistics and stopping rules: The trial will be stopped at any time that there is reasonable evidence that the true rate of day +100 nonrelapse mortality exceeds 0.40. It is the intention to include an initial 20 patients.

DETAILED DESCRIPTION:
PROTOCOL SYNOPSIS

Title of the study A pilot study to assess the feasibility of unrelated umbilical cord blood transplantation with coinfusion of third-party mesenchymal stem cells after myeloablative or nonmyeloablative conditioning in patients with hematological malignancies.

Design of the study This is a multicenter single arm, phase I-II pilot study.

Primary objective The primary objective of this study is to determine the feasibility of UCB HSCT with co-infusion of third party mesenchymal stem cells as assessed by the treatment-related mortality at d100 after transplant.

Secondary objectives

* Chimerism at multiple time points
* Hematopoietic recovery (neutrophil and platelet engraftment)
* Immune recovery
* Incidence of acute and chronic graft-versus-host disease (GVHD)
* Infectious complications
* Disease free survival
* Relapse incidence
* Overall survival

Graft criteria

* No peripheral blood or marrow donor available at the 9/10 compatibility level using high resolution typing techniques
* Adequate cord blood transplant available:

  a)Single cord blood
* Minimal 4/6 match (DR1-high, A-low, B-low)
* Minimal 2 (6/6), 2.5 (5/6) or 3 (4/6) x 10exp7 nucleated cells per kg in the graft b)Double cord blood
* At least 4/6 common antigens shared by recipient and the 2 cord blood transplants
* Minimal 3x 10exp7 nucleated cells per kg in the combined graft

Patient inclusion criteria

* Age 15-60 yrs
* Allogeneic stem cell transplantation is the preferred treatment option:

  a)High risk acute myeloid leukemia (AML) in first complete remission (CR)
* Preceding myelodysplastic syndrome
* High risk karyotypes (e.g. monosomy 5 or 7, complex)
* Feline McDonough Sarcoma (FMS)-like tyrosine kinase 3 (FLT3) alteration
* > 2 cycles to obtain CR
* Erythroblastic or megakaryocytic leukemia b)High risk acute lymphoblastic leukemia (ALL) in first CR
* High risk karyotypes (e.g. t[9;22], t[4;11], t[1;19], complex)
* Mixed lineage leukemia (MLL) rearrangements c)Acute leukemia in second or third remission d)High risk myelodysplastic syndrome: International Prognostic Scoring System (IPSS) Intermediate-2 or high risk e)Advanced lymphoproliferative disorders
* Diffuse large B-cel non-Hodgkin lymphoma (NHL) or mantle cell NHL or B-prolymphocytic leukemia

  * Sensitive relapse after autologous HSCTx
* T-prolymphocytic leukemia
* Chronic lymphocytic leukemia

  * Refractory to fludarabine
  * Adverse karyotypes (del p17) f)Chronic myeloid leukemia
* Refractory or intolerant to second-line tyrosine kinase inhibitors g)Multiple myeloma
* Advanced disease (selected cases)
* Informed consent given

Patient exclusion criteria

* Previous allogeneic transplant
* Progressive malignant disease
* Significant organ damage as a contraindication to allotransplantation

  * Creatinine clearance < 60 ml/min
  * Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) > 3x normal value and/or serum bilirubin >3 mg/dL
  * Cardiac failure (LVEF < 50%)
  * Clinical relevant pulmonary disease: Diffusing capacity of lung for carbon monoxide (DLCO) < 50% normal
* Significant psychiatric or neurological disorder
* Uncontrolled viral, fungal or bacterial infection
* Pregnancy
* HIV positive

Study procedure Patients will receive either myeloablative or reduced intensity conditioning. One or 2 cord blood transplants will be transplanted, followed by infusion of a third-party mesenchymal stem cell transplant

Adverse event reporting BHS transplant committee will establish a protocol review committee which will organize a central monitoring of the study. Within the context of allogeneic HSCTx many severe events are likely to occur.

Statistics and stopping rules The trial will be stopped at any time that there is reasonable evidence that the true rate of day +100 nonrelapse mortality exceeds 0.40. It is the intention to include an initial 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic stem cell transplantation is the preferred treatment option:
* High risk acute myeloid leukemia (AML) in first complete remission (CR)
* Preceding myelodysplastic syndrome
* High risk karyotypes (e.g. monosomy 5 or 7, complex)
* FLT3 alteration
* > 2 cycles to obtain CR
* Erythroblastic or megakaryocytic leukemia
* High risk acute lymphoblastic leukemia (ALL) in first CR
* High risk karyotypes (e.g. t[9;22], t[4;11], t[1;19], complex)
* MLL rearrangements
* Acute leukemia in second or third remission
* High risk myelodysplastic syndrome: IPSS Intermediate-2 or high risk
* Advanced lymphoproliferative disorders
* Diffuse large B-cel non-Hodgkin lymphoma (NHL) or mantle cell NHL or
* B-prolymphocytic leukemia
* Sensitive relapse after autologous HSCTx
* T-prolymphocytic leukemia
* Chronic lymphocytic leukemia
* Refractory to fludarabine
* Adverse karyotypes (del p17)
* Chronic myeloid leukemia
* Refractory or intolerant to second-line tyrosine kinase inhibitors
* Multiple myeloma
* Advanced disease (selected cases)
* Informed consent given

Exclusion Criteria:

* Previous allogeneic transplant
* Progressive malignant disease
* Significant organ damage as a contraindication to allotransplantation
* Creatinine clearance < 60 ml/min
* AST/ALT > 3x normal value and/or serum bilirubin > 3 mg/dL
* Cardiac failure (LVEF < 50%)
* Clinical relevant pulmonary disease: DLCO < 50% normal
* Significant psychiatric or neurological disorder
* Uncontrolled viral, fungal or bacterial infection
* Pregnancy
* HIV positive

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2010-11; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
treatment-related mortality | day 100 after transplant
  death related to treatment procedures

SECONDARY OUTCOMES:
Hematopoietic recovery | One year after transplant
  recovery of peripheral blood counts

CONTACTS AND LOCATIONS:
Overall Officials: Rik Schots, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium